CLINICAL TRIAL: NCT06207578
Title: Long Term Stability of Implants Placed With Crestal Sinus Approach Versus Osseodensification in Atrophic Posterior Maxilla. A Randomized Clinical Trial.
Brief Title: Implants Placed With Crestal Sinus Approach Versus Osseodensification in Atrophic Posterior Maxilla
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, Clinical director of implant speciality program, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDCE.N7
Record Dates: First submitted 2023-12-17; First posted 2024-01-17 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Implants
Keywords: osseodensification; densah bur; Crestal implant approach; closed sinus elevation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implant placement using crestal sinus approach (Experimental): Drilling will be done gently till reaching 0-1mm from the sinus floor, then implant placement will take place and the implant itself will be used to gently elevate the sinus up to 3-5mm.
  Interventions: Procedure: implant placement using crestal sinus approach
- Implant placement using osseodensification (Active Comparator): Using Densah bur kit foe osteotomy preparation followed by implant placement
  Interventions: Procedure: Implant placement using osseodensification

INTERVENTIONS:
Procedure: implant placement using crestal sinus approach — a Full thickness flap will be elevated at the edentulous site with two vertical releasing incision. After flap reflection, the preparation of osteotomy will be prepared following standard implant system protocol preparation of the osteotomy. Drilling will be done gently till reaching 0-1mm from the sinus floor, then implant placement will take place and the implant itself will be used to gently elevate the sinus up to 3-5mm
  Arms: Implant placement using crestal sinus approach
Procedure: Implant placement using osseodensification — The implant motor will be adjusted on reverse mode with 800 to 1200 rpm. According to the desired implant dimension, Densah bur diameter will be used and then implant placement.
  Arms: Implant placement using osseodensification

SUMMARY:
However, recently, most described techniques for posterior atrophic maxillary rehabilitation, are targeting more conservative, cost-effective and efficient methods for sinus elevation eliminating its lateral access. The aim of the present study is to evaluate and compare the long-term implant stability for implants placed by the novel crestal sinus approach versus osseodensification using Densa-bur in Atrophic Posterior Maxilla.

DETAILED DESCRIPTION:
Rehabilitation of the edentulous posterior maxilla using osseointegrated implants is often challenging due alveolar bone resorption, low bone density and maxillary sinus pneumatization. Many protocols were suggested to overcome this phenomenon; placing short implants, 2nd premolar occlusion and finally maxillary sinus elevation.

Maxillary sinus elevation is one of the most common surgical techniques used for increasing the available bone volume to place implants and restore function and esthetics. Sinus elevation was introduced when Boyne and James presented lateral window approach as a modification of the Coldwell Luc technique; the access to lift the sinus floor is performed by a window through the lateral wall. This technique was proven to be effective and successful for sinus elevation even up to 12 mm in cases of severely atrophic ridge. It was later divided into three techniques according to the lateral wall preparation; hinge, elevated and complete.

Lateral approach for sinus lift is usually indicated when residual bone height is less than 5mm. While transcrestal approach can be successfully adopted when residual bone height is at least 5 mm. Osteotome sinus floor elevation was 1st introduced by Summers (1994) and proved to be less invasive, more conservative, less time consuming, and reduces postoperative discomfort to the patient.

Osseodensification is a new surgical technique of biomechanical bone preparation performed for dental implant placement where bone is compacted and autografted into open marrow spaces and osteotomy site walls in outwardly expanding directions. The use of densah burs for preparing implant site had many advantages including the increase of implant bone contact by compaction autografting rather than excavation of bone in conventional drill, this mainly depends on the viscoelastic nature of bone where time dependent stress produces time dependent strain, it also allows for higher insertion torque and increased stability of dental implant.

The use of densah burs for maxillary sinus lifting was first introduced by Huwais and Meyer utilizing the advantages of the osseodensification approach for elevation of the maxillary sinus floor. The idea of compaction autografting supported by the design of densah burs with specially tapered geometry and specially designed flutes to compact the bone on its walls and apex. The idea of this concept is that the special design of flutes in the densifying non cutting mood with counter clockwise motion and presence of irrigation cause a hydraulic wave at the apex of the bur, this wave cause pushing of the sinus membrane upward, also in presence of grafting material cause the same effect and subsequent elevation of the Schneiderian membranewith limited risk of perforation. So this approach is suggested to provide a safe technique for maxillary sinus lifting with limited complications as in osteotome or lateral approach, less perforation and less invasiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Edentulous atrophic posterior maxillary ridge.
2. Residual alveolar ridge height within 5-6 mm.
3. At least 2mm band of keratinized tissue.
4. Patients with good oral hygiene.
5. Compliant patients to the follow up periods.

Exclusion Criteria:

1. Medically compromised patients.
2. Smokers.
3. Pregnant females.
4. Patients with active periodontal disease.
5. Bruxer patients.
6. Patients with chronic or active sinusitis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Long- term Implant Stability | 12 months
  Resonance frequency analysis will be employed with a dedicated device (Osstell). For each implant, implant stability quotient ISQ values will measured from the four sites (mesial, distal, buccal, and palatal sites). The mean of all measurements will be rounded to a whole number and regarded as the final ISQ of the implant. ISQ values will obtained after implant placement (T1), after loading (T2), 6 months after loading (T3) follow up intervals.

SECONDARY OUTCOMES:
Implant survivability | 12 months
  Individual unattached implant that is immobile when tested clinically, radiography that does not demonstrate evidence of peri-implant radiolucency, Bone loss that is less than 0.2 mm annually after the implant's first year of service, No persistent pain, discomfort or infection
Vertical bone height formed | 12 months
  using CBCTs 1
Post operative pain | 10 days
  will be recorded by the patient for 10 days after the surgery The patients will mark the pain perception in a non-numerical 100 mm line ranging from "no pain=0" (left) to "very painful=100" (right). It will be given a numerical value by measuring in millimeters the distance from the left end of the line

IPD SHARING:
Plan to Share IPD: No